CLINICAL TRIAL: NCT02224326
Title: Prospective Study to Evaluate the Predictive Value of Vagus Somatosensory Evoked Potentials (VSEP) and Near-infrared Spectroscopy (NIRS) in the Early Diagnosis of Alzheimer´s Disease
Brief Title: Vagus Somatosensory Evoked Potentials and Near-infrared Spectroscopy in the Early Diagnosis of Dementia
Acronym: Vogel
Status: Completed | Type: Observational
Sponsor: University of Wuerzburg (Other)
Responsible Party: Principal Investigator, Thomas Polak, Senior Physician, University of Wuerzburg
Other Study IDs: Vogel-1
Record Dates: First submitted 2013-09-07; First posted 2014-08-25 (Estimated); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Alzheimer´s Disease
Keywords: Alzheimer´s disease; early diagnosis; evoked potentials; near-infrared spectroscopy
MeSH Terms: conditions — Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood, serum
Oversight: Data Monitoring Committee: No

SUMMARY:
In its long preclinical course, AD shows a spreading pattern of specific pathology in a uniform sequence of predictable steps including brainstem nuclei in early stages. Many of these nuclei which are early involved in AD take equally part in the afferences of the Xth cranial nerve, the Vagus nerve. A method for the functional assessment of Vagus-related nuclei in the lower brainstem is the technique of somatosensory evoked potentials of the Vagus nerve (VSEP). This method targets the accessibility of early functional changes by evoked potentials on one hand and the early affection of specific brainstem nuclei comprising Vagus afferences in the course of AD on the other hand. The method of VSEP takes advantage of the transcutaneous stimulation of the auricular branch of the Vagus nerve (ABVN) which is presumed to be the only sensory part of this nerve innervating parts of the outer meatus acoustics at the tragus. This cutaneous branch was shown to gain access to Vagus afferences via brainstem regions which are affected in the course of AD. VSEP latencies in AD were shown to be significantly longer as compared to healthy controls. Yet, if VSEP really are suited for the early detection of AD is still not known.

Functional near-infrared spectroscopy (fNIRS) measures changes in cerebral oxygenation by means of near-infrared light using wavelengths of 650-850 nm. The principle of fNIRS is based on the principle that regional neuronal activation of the brain leads to an increase in metabolism and oxygenation of brain tissue in that region which is accompanied by an elevated regional cerebral blood flow. In AD, there is a growing body of literature reporting deviant fNIRS activation patterns for a variety of tasks. For example, it was shown that the fNIRS activation pattern in frontal and parietal cortex areas in subjects with AD performing the line orientation paradigm is clearly different from healthy controls. Yet, if fNIRS is suited as a means of early detection of AD is not known.

Therefore we aimed at testing the predictive value of VSEP and fNIRS in the early detection of AD. The hypothesis to be tested within this study states that subjects developing AD or MCI within an observation period of 6 years depict longer VSEP latencies, a different fNIRS oxygenation pattern and a lower performance in neuropsychologic rating below the level of dementia at baseline than those who remain cognitively stable.

DETAILED DESCRIPTION:
With the increasing life span of our population, the prevalence of dementia syndromes is increasing. The most frequent cause of dementia is Alzheimer´s disease (AD), and still, it is not curable. Thus, AD is of increasing medical, social and economic importance.

Intensive scientific work within the past 30 years has identified a range of different factors contributing to the pathogenesis of AD. These complex processes result in specific therapeutic options which are currently investigated in clinical trials. Regardless of the considered risk factor or the specific therapeutic intervention, treatment should be started as early in the excessive preclinical process of AD as possible since it can interfere with the formation of amyloid plaques or neurofibrils. Especially neuroprotective interventions are more effective the less neurons are irreversibly damaged.Therefore, an early diagnosis of developing or incipient AD should be of utmost importance. Likewise, in the light of therapeutic options specific for AD, its differential diagnosis from other forms of dementia seems important.

Therefore, an ideal examination method should not only be easy to conduct, cost effective, repeatable, non-invasive and without discomfort for patients, but it should in particular detect early stages of disease and it should, if possible, consider the development of AD-specific changes. Obviously, today´s routine examination methods in the diagnosis of AD or MCI such as magnetic resonance imaging, cerebrospinal fluid analysis or positron emission tomography do not fulfil all of these requirements. Thus, in the absence of a single diagnostic test and realizing the necessity to combine biomarkers to increase the diagnostic accuracy there is still need for methods that circumvent all those disadvantages.

Since early cellular changes of the disease are expected to impact brain function long before severe morphological alterations occur, these changes should primarily be investigated using functional examination which can be conducted with neurocognitive methods such as intensive neuropsychological rating or with electrophysiological or functional brain imaging methods.

Neuropsychological rating Prior studies investigated the predictive validity of different cognitive measures for the development of AD such as associative learning, verbal fluency and constructive praxis. As such, verbal and non-verbal memory, visual-spatial and executive functions and verbal fluency with executive component seem to be suited for following the deterioration of cognition. In subjects who later develop AD or MCI as compared to a healthy controls, worse performance in episodic memory according (Delayed Verbal and Visual Memory und Associative Learning) and in semantic verbal fluency are known to be characteristic. An extended neuropsychologic testing to measure these cognitive processes thus seems reasonable in particular to evaluate the additional benefit of other diagnostic methods.

Vagus somatosensory evoked potentials (VSEP) As we know today, AD has a long preclinical course with a spreading pattern of specific AD pathology such as neurofibrillary tangles in a uniform sequence of predictable steps. Many of these nuclei which are early involved in AD like the Locus caeruleus, parabrachial nucleus or Raphe nuclei take equally part in the afferences of the Xth cranial nerve, the Vagus nerve. Our laboratory used a hypothesis-driven approach to develop a method for the functional assessment of Vagus-related nuclei in the lower brainstem which resulted in the technique of somatosensory evoked potentials of the Vagus nerve (VSEP). This method targets the accessibility of early functional changes by evoked potentials on one hand and the early affection of specific brainstem nuclei comprising Vagus afferences in the course of AD on the other hand.

The method of VSEP takes advantage of the transcutaneous stimulation of the auricular branch of the Vagus nerve (ABVN). It is presumed to be the only sensory part of this nerve innervating parts of the outer meatus acoustics at the tragus. This cutaneous branch was shown to gain access to Vagus afferences via the Solitary tract nucleus which is affected in the course of AD as well.

The technique of VSEP meanwhile is well characterized from a methodological point of view. There are numerous findings suggesting that observed potentials are generated at brainstem level and can be detected as far field potentials at the scalp without any side effects. VSEP are reproducible and amplitudes as well as latencies are in the range of corresponding parameters of acoustic evoked potentials. Detailed examinations with functional magnetic imaging revealed a cortical activation pattern upon ABVN stimulation comparable to the activation pattern as response to the conventional invasive stimulation of the main Vagus branch. In a subsequent work, even involvement of brainstem activation was demonstrated that could be related to ascending Vagus nerve projections.

As such, VSEP were proposed as a possible means for the early detection of AD and mild cognitive impairment (MCI). VSEP latencies in both groups were shown to be significantly longer as compared to healthy controls. No difference in VSEP parameters was found in patients with Vascular dementia and Major depression.

Near-infrared spectroscopy (NIRS) NIRS measures changes in cerebral oxygenation by means of near-infrared light using wavelengths of 650-850 nm. The principle of NIRS is based on the principle of neurovascular coupling stating that regional neuronal activation of the brain leads to an increase in metabolism and oxygenation of brain tissue in that region which is accompanied by an elevated regional cerebral blood flow. This in turn leads to an increased oxygen saturation with elevated concentrations of oxygenated haemoglobin and diminished concentrations of deoxygenated haemoglobin.

In the last years, functional NIRS (fNIRS) was increasingly applied to measure changes in oxygen saturation of cortical areas during a variety of cognitive tasks such as for example verbal fluency test and thus to detect specific cortical activation not only in the visual and the motor system, but also in cortical areas relevant for cognitive tasks such as prefrontal and parietal cortex that remain stable and are replicable. In AD, there is a growing body of literature reporting deviant fNIRS activation patterns for a variety of tasks. For example, young healthy subjects displayed a distinct activation pattern of the prefrontal cortex during a verbal fluency test (VFT) showing a left hemispheric lateralization which decreased with age without a decline in behavioural performance. In contrast, subjects with AD showed a worse behavioural performance and an even more severe decrease of prefrontal activation as well as a reduced left lateralization as compared to an age-adjusted healthy control group. Likewise, it was shown that the fNIRS activation pattern in frontal and parietal cortex areas in subjects with AD performing the line orientation paradigm is clearly different from healthy controls.

Aim of the study To summarize, VSEP, fNIRS and neuropsychological rating are able to differentiate AD from healthy controls. From a theoretical point of view, these methods should even be suited as a means of detection of the disease in early phases as well. If they are really suited as means for that purpose is to be examined in the here presented study. Therefore we aimed at testing the predictive value of these methods in the early detection of AD. In the here presented research project, 600 subjects examined at baseline by means of VSEP, fNIRS and extended neuropsychological, somatic and laboratory examination are to be reexamined 3 and 6 years later. The hypothesis to be tested within this study states that subjects developing AD or MCI within the observation period depict longer VSEP latencies, a different fNIRS oxygenation pattern and a lower performance in neuropsychologic rating below the level of dementia at baseline than those who remain cognitively stable.

ELIGIBILITY:
Inclusion Criteria:

* inhabitant of Wuerzburg
* born between 1.4.1936 and 31.3.1941
* able to give informed consent

Exclusion Criteria:

* manifestation of - apart from dementia - other severe psychiatric disease such as Schizophrenia, neurologic disease such as Parkinson´s disease or stroke or intern disease such as cancer within the past 12 months
* severe, uncorrected see or hearing disturbance

Ages: 70 Years to 78 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Inhabitants of Wuerzburg, the 130 000 inhabitants capital of the german district Lower Franconia who are born between 1.4.1936 and 31.3.1941
Sampling Method: Non-Probability Sample
Enrollment: 604 (Actual)
Dates: Start 2011-06; Primary Completion 2023-01 (Actual); Study Completion 2023-01 (Actual)

PRIMARY OUTCOMES:
Mini Mental State Examination (MMSE) | 6 years

SECONDARY OUTCOMES:
Dementia detection test | 6 years

OTHER OUTCOMES:
Activities of daily living scale | 6 years

CONTACTS AND LOCATIONS:
Overall Officials: Jürgen Deckert, MD, Principal Investigator — University Clinic Wuerzburg, Dept. of Psychiatry, Psychosomatics and Psychotherapy, Fuechsleinstrasse 15, D-97080 Wuerzburg, Germany; Thomas Polak, MD, Study Director — University Clinic Wuerzburg and Hephata Diakonie, Hauptstraße 280, D-63879 Weibersbrunn, Germany; Martin J Herrmann, PhD, Study Director — University Clinic Wuerzburg, Dept. of Psychiatry, Psychosomatics and Psychotherapy, Fuechsleinstrasse 15, D-97080 Wuerzburg, Germany; Martin Lauer, MD, Study Director — University Clinic Wuerzburg, Dept. of Psychiatry, Psychosomatics and Psychotherapy, Fuechsleinstrasse 15, D-97080 Wuerzburg, Germany
Locations (1):
- University Clinic Wuerzburg, Würzburg, Germany

REFERENCES:
- [Background] Katzorke A, Zeller JBM, Muller LD, Lauer M, Polak T, Deckert J, Herrmann MJ. Decreased hemodynamic response in inferior frontotemporal regions in elderly with mild cognitive impairment. Psychiatry Res Neuroimaging. 2018 Apr 30;274:11-18. doi: 10.1016/j.pscychresns.2018.02.003. Epub 2018 Feb 11. PMID 29472145
- [Background] Zeller JBM, Katzorke A, Muller LD, Breunig J, Haeussinger FB, Deckert J, Warrings B, Lauer M, Polak T, Herrmann MJ. Reduced spontaneous low frequency oscillations as measured with functional near-infrared spectroscopy in mild cognitive impairment. Brain Imaging Behav. 2019 Feb;13(1):283-292. doi: 10.1007/s11682-018-9827-y. PMID 29362991
- [Background] Polak T, Herrmann MJ, Muller LD, Zeller JBM, Katzorke A, Fischer M, Spielmann F, Weinmann E, Hommers L, Lauer M, Fallgatter AJ, Deckert J. Near-infrared spectroscopy (NIRS) and vagus somatosensory evoked potentials (VSEP) in the early diagnosis of Alzheimer's disease: rationale, design, methods, and first baseline data of the Vogel study. J Neural Transm (Vienna). 2017 Nov;124(11):1473-1488. doi: 10.1007/s00702-017-1781-0. Epub 2017 Sep 1. PMID 28864837
- [Derived] Herrmann MJ, Wuttke A, Breuninger L, Eff J, Ettlinger S, Fischer M, Gotzelmann A, Gram A, Pomper LD, Schneider E, Schwitalla L, Siminski N, Spielmann F, Weinmann E, Weyel V, Zeller JBM, Lauer M, Deckert J, Polak T. Functional near-infrared spectroscopy and vagus somatosensory evoked potentials add to the power of established parameters such as poor cognitive performance, dsyosmia and APOe genotype to predict cognitive decline over 8 years in the elderly. J Neural Transm (Vienna). 2025 Mar;132(3):455-468. doi: 10.1007/s00702-024-02859-y. Epub 2024 Nov 13. PMID 39535568